CLINICAL TRIAL: NCT05516589
Title: Neoadjuvant Chemotherapy, Tislelizumab With Afatinib for the Treatment of Resectable Head and Neck Squamous Cell Carcinoma: A Single-Arm Phase 2 Trial (neoCHANCE-2 Trial)
Brief Title: Neoadjuvant Chemotherapy, Tislelizumab With Afatinib for HNSCC
Acronym: neoCHANCE-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiECRCT20210621
Record Dates: First submitted 2022-08-19; First posted 2022-08-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; Neoadjuvant therapy; Immunotherapy; EGFR-TKI; Chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Cisplatin; tislelizumab; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): Participants will receive
  * TP chemotherapy every 3 weeks x 2 cycles (Nab-paclitaxel 260mg/m^2 IV on day1, Cisplatin 75mg/m^2 IV on day 1);
  * Tislelizumab 200mg IV every 3 weeks x 2 cycles;
  * Afatinib 30mg PO everyday x 6 weeks.
  Interventions: Drug: Nab-paclitaxel; Drug: Cisplatin; Biological: Tislelizumab; Drug: Afatinib

INTERVENTIONS:
Drug: Nab-paclitaxel — 260mg/m^2 IV Q3W
  Other Names: Albumin-bound paclitaxel; Abraxane
Drug: Cisplatin — 75mg/m^2 IV Q3W
  Other Names: CDDP
Biological: Tislelizumab — 200mg IV Q3W
  Other Names: BGB-A317
Drug: Afatinib — 30mg PO QD

SUMMARY:
To explore the efficiency and safety of TP chemotherapy, tislelizumab, combined with afatinib as a new neoadjuvant treatment regimen for patients with resectable HNSCC.

DETAILED DESCRIPTION:
More than 60% of patients with Head and neck squamous cell carcinoma (HNSCC) have locally advanced or metastatic disease at the time of diagnosis, with a 5-year overall survival rate of less than 60%. The clinical outcomes of those patients still need to be improved.

Neoadjuvant therapy theoretically could reduce tumor volume, increase organ retention rate, and improve clinical prognosis. However, results from several phase III clinical trials have not proved a significant survival benefit of neoadjuvant chemotherapy for patients with resectable HNSCC except for nasopharyngeal carcinoma. There is an urgent need to explore new neoadjuvant treatment options for those patients.

Immunotherapy such as PD-1/PD-L1 inhibitors have shown excellent efficiency in the treatment of malignancies. Anti-PD-1 therapy is approved as the first-line treatment of recurrent/metastatic HNSCC. Neoadjuvant immunotherapy for the treatment of locally advanced and resectable HNSCC has been demonstrated to be feasible in some trials.

Afatinib, as an irreversible ErbB tyrosine kinase inhibitor (TKI), has been used as the second-line treatment for recurrent and/or metastatic HNSCC. A previous study published in 2018 confirmed that afatinib can be administered safely before surgery.

In summary, we designed this study to explore the efficiency and safety of chemotherapy (TP regimen), anti-PD1 immunotherapy (tislelizumab), combined with EGFR-TKI (afatinib) as a new neoadjuvant treatment regimen for patients with resectable HNSCC, aiming to provide a new treatment option for those patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above.
2. Patients with pathologically confirmed HNSCC (except for nasopharyngeal carcinoma) and meet the following conditions:

   * were newly diagnosed and without distant metastasis;
   * were deemed surgically resectable evaluated by a head and neck surgeon;
   * were willing to undergo surgery.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
4. Adequate organ and bone marrow function:

   * absolute neutrophil count ≥ 1.5 × 10^9/L, hemoglobin ≥ 80 g/L, platelets ≥ 80 × 10^9/L;
   * ALT, AST and ALP < 2.5× upper limit of normal (ULN), total bilirubin ≤ 2×ULN;
   * albumin≥ 2.8 g/dL；
   * creatinine clearance ≥ 60 ml/min；
   * INR≤ 1.5；APTT≤ 1.5×ULN；
5. Written informed consent.

Exclusion Criteria:

1. History of other malignancies (except for the history of malignant tumors that have been cured and have not recurred within 5 years, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, in situ cervical cancer, and gastrointestinal mucosal cancer, etc.）
2. Have an active autoimmune disease requiring systemic treatment or a documented history of clinically severe autoimmune disease.
3. Any history of allergic disease, or a sever hypersensitivity reaction to drugs, or allergy to the study drug components.
4. Any of prior therapy with:

   * anti-PD-1, anti-PD-L1/2, anti-CTLA-4 antibody, anti-EGFR antibody or EGFR-TKIs；
   * antitumor vaccine;
   * any active vaccine against an infectious disease within 4 weeks prior to the first dose or planned during the study period;
   * major surgery or serious trauma within 4 weeks before the first dose;
   * toxicity from prior antitumor therapy has not recovered to ≤ CTCAE Version 5.0 Grade 1 or the level specified by the inclusion/exclusion criteria.
5. With serious medical diseases, such as grade II and above cardiac dysfunction (NYHA criteria), ischemic heart disease, supraventricular or ventricular arrhythmia, poorly controlled diabetes mellitus, poorly controlled hypertension, echocardiographic ejection fraction < 50%, etc.
6. With interstitial pneumonitis, non-infectious pneumonitis, active pulmonary tuberculosis, or history of pulmonary tuberculosis infection that were not controlled by treatment.
7. With hyperthyroidism, or organic thyroid disease.
8. With active infection, or unexplained fever during the screening period or 48 hours before the first dose.
9. With active hepatitis B or C, or known history of positive HIV test, or acquired immunodeficiency syndrome.
10. History of a clear neurological or psychiatric disorder.
11. History of drug abuse or alcohol abuse.
12. Women who are pregnant or breastfeeding, or have a reproductive plan from the screening period to 3 months after the end of the study, or have sex without contraceptive measures, or are unwilling to take appropriate contraceptive measures.
13. Received any investigational drug within 4 weeks prior to the first dose, or concurrently enrolled in another clinical trial.
14. Any other factors that are not suitable for inclusion in this study judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pathologic Complete Response | Time of surgery
  Pathologic complete response was defined as the absence of viable tumor cells.

SECONDARY OUTCOMES:
Major Pathologic Response | Time of surgery
  Major pathologic response was defined as fewer than 10% viable tumor cells.
Objective Response Rate | Up to 8 weeks
  Objective response rate was defined as the percentage of participants with a best overall response of CR or PR using RECIST Criteria
Adverse Events | Up to 12 weeks
  Adverse events included adverse events using CTCAE Criteria and unplanned surgery delays.
Disease-free Survival | 1 year
  Disease-free survival was defined as the time from the administration of the first dose to first disease progression or death.
Overall Survival | 1 year
  Overall survival was defined as the time from the administration of the first dose to death.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Professor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China